CLINICAL TRIAL: NCT01382732
Title: Carbetocin Versus Oxytocin for Prevention of Postpartum Hemorrhage in Patients With Severe Preeclampsia: a Double Blind Randomized Controlled Trial
Brief Title: Carbetocin vs. Oxytocin for Prevention of Postpartum Bleeding in Patients With Severe Preeclampsia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., MD, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MHST2011-06
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Severe Preeclampsia; Postpartum Hemorrhage
Keywords: Pre-eclampsia; Postpartum hemorrhage; Carbetocin; Oxytocin
MeSH Terms: conditions — Pre-Eclampsia; Postpartum Hemorrhage | interventions — carbetocin; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carbetocin (Experimental): Protocol A (carbetocin + placebo) Carbetocin: 100ug (1mL) + Ringer's Lactate 10mL directly into the vein in no less than two minutes.
  Ringer's Lactate 4mL applied to a bag with 1000mL of Ringer's Lactate to be passed intravenously at a rate of 125mL/hr
  Interventions: Drug: Carbetocin
- Oxytocin (Active Comparator): Protocol B (oxytocin + placebo) Ringer's Lactate 11mL directly into the vein in no less than two minutes. Oxytocin 20 U (4mL) diluted in a bag with 1000mL of Ringer's Lactate to be passed intravenously at a rate of 125mL/hr
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Carbetocin — Protocol A (carbetocin + placebo) Carbetocin: 100ug (1mL) + Ringer's Lactate 10mL directly into the vein in no less than two minutes.
  Other Names: Lonactene
  Arms: Carbetocin
Drug: Oxytocin — Oxytocin 20 U (4mL) diluted in a bag with 1000mL of Ringer's Lactate to be passed intravenously at a rate of 125mL/hr
  Other Names: Pitocin
  Arms: Oxytocin

SUMMARY:
Postpartum hemorrhage is an important cause of maternal morbidity and mortality. In patients with severe preeclampsia there is an increased risk of postpartum hemorrhage but the hemodynamic changes associated with this pathology make the management of any kind of bleeding particularly troublesome. There are many pharmacological options, being oxytocin the first line of treatment. However there is no evidence about the safety and efficacy of carbetocin, an oxytocin agonist. The investigators aimed to compare oxytocin with carbetocin for the routine prevention of postpartum hemorrhage in patients with severe preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 28 weeks and term
* Severe pre-eclampsia

Exclusion Criteria:

* Twin pregnancy
* Coagulation disorders
* HELLP Syndrome
* Eclampsia

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 636 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Need for additional uterotonics | Six months
  Number of cases allocated to one arm of the study that due to the presence of continous bleeding postpartum need the use of an additional uterotonic.

SECONDARY OUTCOMES:
Development of oliguria | six months
  Number of cases that develop oliguria (<30 mL/hr over a 2 hour period) after the administration of the drug.
Changes in hemodynamic status | six months
  Changes in Systolic pressure , dyastolic pressure, mean arterial pressure and heart rate one and two hours after the administration of the drug.

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo A Reyes, MD, Principal Investigator — Saint Thomas Hospital, Panama
Locations (1):
- Saint Thomas H, Panama City, Provincia de Panamá, Panama